CLINICAL TRIAL: NCT03270163
Title: Evaluation of Muscle Strength by Transcutaneous Electrical Stimulation in Intensive Care Unit Patients
Brief Title: Evaluation of Muscle Strength by Transcutaneous Electrical Stimulation
Acronym: STRENGTH-ICU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no more inclusions possible
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Laboratoire de Physiologie de l'Exercice (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1708055; 2017-A00919-44 (Other: ANSM)
Record Dates: First submitted 2017-08-10; First posted 2017-09-01 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Muscle Weakness
Keywords: Intensive care unit acquired muscle weakness; Transcutaneous electrical stimulation; magnetic stimulation
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Magnetic and Transcutaneous electrical stimulation of quadriceps
  Interventions: Diagnostic Test: Transcutaneous electrical stimulation; Diagnostic Test: Magnetic stimulation; Diagnostic Test: ultrasound measurement

INTERVENTIONS:
Diagnostic Test: Transcutaneous electrical stimulation — The following tests and measurements will be carried out on the patient within 3 days of inclusion and again between the 4th and 6th day after inclusion and upon awakening:
  * three simple electrical stimulations,
  * three electrical doublets at the frequency of 100Hz
  For each type of electrical stimulation, the stimulations will be carried out 3 times and reproduced at 1 hour intervals.
Diagnostic Test: Magnetic stimulation — The following tests and measurements will be carried out on the patient within 3 days of inclusion and again between the 4th and 6th day after inclusion and upon awakening:
  * three simple magnetic stimulations,
  * three magnetic doublets at the frequency of 100Hz
  For each type of magnetic stimulation, the stimulations will be carried out 3 times and reproduced at 1 hour intervals.
Diagnostic Test: ultrasound measurement — The ultrasound measurement of the thickness of the quadriceps muscle will be carried out on the patient within 3 days of inclusion and again between the 4th and 6th day after inclusion and upon awakening.

SUMMARY:
Acquired Neuromyopathy of Resuscitation (NMAR) is a common condition. Its diagnosis is difficult and often late because it is based on a clinical assessment of muscle strength (MRC score) requiring the patient to be awake and cooperative.

Transcutaneous electrical stimulation consists of applying electrical stimulation along the path of a motor nerve in order to generate contraction of the previously relaxed muscle. The mechanical response thus generated is recorded and allows the muscular strength developed to be assessed. Non-invasive and easily performed in the patient's bed, transcutaneous electrical stimulation could be an interesting alternative for early assessment of muscle strength in the still sedated resuscitation patient. However, this technique could be perceived as uncomfortable or painful in the awake patient so that magnetic stimulation, which is generally much better tolerated, should be preferred. However, magnetic stimulators have a limited maximum magnetic field which may prevent supramaximal stimulation especially in patients developing generalized edema (i.e., in the initial resuscitation phase).

DETAILED DESCRIPTION:
We propose to conduct a reproducibility study of quadriceps force measurement in patients undergoing resuscitation by transcutaneous electrical and/or magnetic neurostimulation in the initial (i.e., < 96 h) and late (> 96 h) phases of resuscitation and then in the recovery phase. For each investigative technique (i.e., electrical vs. magnetic), we will perform 2 types of stimulation: single stimulation and high frequency doublet stimulation (100 Hz), repeated 3 times each.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* admitted in intensive care unit B of ST-Etienne hospital
* Predictable duration of mechanical ventilation of more than 72 hours
* Patient whose family has given informed and written consent to the patient's participation in the study

Exclusion Criteria:

* Pregnant woman,
* Patients with peripheral nerve damage prior to or at the time of measurement
* Curarized patients (non-efficacy of neurostimulation)
* Fracture of limb or pelvis
* Presence of a catheter in the stimulation zone (femoral artery or vein)
* Patients suffering from psychiatric pathologies.
* Brain pathology leading the patient to intensive care.
* Patients with neuromuscular pathology.
* Patients carrying equipment subject to possible electrical and/or magnetic interference,
* Patient with spinal fracture(s) at risk of spinal cord injury

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Reproductibility | At day 2
  Reproductibility of the force measurement after electrical muscle stimulation by a doublet at 100 Hz.

SECONDARY OUTCOMES:
Reproductibility | At day 4
  Reproductibility of the force measurement after electrical muscle stimulation by a doublet at 100 Hz.
Reproductibility | when the patient wakes up (on average 15 days)
  Reproductibility of the force measurement after electrical muscle stimulation by a doublet at 100 Hz.
Reproductibility | At day 2
  Reproductibility of the force measurement after magnetic muscle stimulation by a doublet at 100 Hz.
Reproductibility | At day 4
  Reproductibility of the force measurement after magnetic muscle stimulation by a doublet at 100 Hz.
Reproductibility | when the patient wakes up (on average 15 days)
  Reproductibility of the force measurement after magnetic muscle stimulation by a doublet at 100 Hz.
Reproductibility | At day 2
  Reproductibility of the force measurement after one simple electrical muscle stimulation
Reproductibility | At day 4
  Reproductibility of the force measurement after one simple electrical muscle stimulation
Reproductibility | when the patient wakes up (on average 15 days)
  Reproductibility of the force measurement after one simple electrical muscle stimulation
Reproductibility | At day 2
  Reproductibility of the force measurement after one simple magnetic muscle stimulation
Reproductibility | At day 4
  Reproductibility of the force measurement after one simple magnetic muscle stimulation
Reproductibility | At day 6
  Reproductibility of the force measurement after one simple magnetic muscle stimulation
Intensive care unit acquired muscle weakness (ICUAW) | 1 month
  Occurrence of ICUAW defined by a MRC score less than 48

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme MOREL, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No